CLINICAL TRIAL: NCT01732770
Title: A Randomized Double-blind Study to Evaluate the Safety and Efficacy of Denosumab Compared With Zoledronic Acid in Postmenopausal Women With Osteoporosis Previously Treated With Oral Bisphosphonates
Brief Title: Safety and Efficacy Study to Evaluate Denosumab Compared With Zoledronic Acid in Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20110153; 2012-001821-28 (EudraCT Number)
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Post Menopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab; Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Denosumab 60 mg (Experimental): Participants received denosumab 60 mg subcutaneous injection once every 6 months for 12 months and placebo to zoledronic acid by intravenous infusion on Day 1.
  Interventions: Biological: Denosumab; Drug: Placebo to Zoledronic Acid
- Zoledronic Acid 5 mg (Active Comparator): Participants received zoledronic acid 5 mg by intravenous infusion on Day 1 and placebo to denosumab by subcutaneous injection on Day 1 and at Month 6.
  Interventions: Drug: Zoledronic Acid; Drug: Placebo to Denosumab

INTERVENTIONS:
Biological: Denosumab — Denosumab 60 mg administered by subcutaneous injection once every 6 months.
  Other Names: Prolia®; AMG 162
  Arms: Denosumab 60 mg
Drug: Zoledronic Acid — Zoledronic acid 5 mg administered by intravenous infusion once a year
  Other Names: Reclast; Aclasta
  Arms: Zoledronic Acid 5 mg
Drug: Placebo to Denosumab — Administered by subcutaneous injection once every 6 months
  Arms: Zoledronic Acid 5 mg
Drug: Placebo to Zoledronic Acid — Administered by intravenous infusion once a year
  Arms: Denosumab 60 mg

SUMMARY:
This study will compare the effectiveness of denosumab treatment every 6 months with once yearly zoledronic acid treatment on bone mineral density (BMD) at various skeletal sites.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory postmenopausal women.
* Age 55 years or older
* Subject has provided informed consent prior to any study specific procedures
* Received oral bisphosphonate therapy for osteoporosis at least 2 years prior to screening visit
* Screening BMD (g/cm²) values at the lumbar spine, total hip or femoral neck values of equal to or less than those listed in the protocol.
* At least 2 lumbar vertebrae and one hip must be evaluable by dual energy x-ray absorptiometry (DXA) at the screening visit

Exclusion Criteria:

* Received other osteoporosis treatment or bone active treatment
* Evidence of history of any of the following:

  * hyperthyroidism (stable on antithyroid therapy is allowed)
  * hypothyroidism (stable on thyroid replacement therapy is allowed)
  * hypo- or hyperparathyroidism
  * hypo- or hypercalcemia based on the central laboratory reference ranges
  * Recent tooth extraction (within 6 months of screening visit)
  * Paget disease of bone (subject report or chart review)
  * other bone diseases which affect bone metabolism (eg, osteopetrosis, osteogenesis imperfecta) (chart review)
* Abnormalities of the following per central laboratory reference ranges:

  * vitamin D deficiency (25[OH] vitamin D level < 20 ng/mL), repletion will be allowed and subjects may be re-screened
  * hypercalcemia
  * elevated transaminases ≥ 2.0 x upper limits of normal (ULN)
* History of any solid organ or bone marrow transplant
* Malignancy (except nonmelanoma skin cancers, cervical or breast ductal carcinoma in situ) within the last 5 years
* Known intolerance to calcium or vitamin D supplements
* Self-reported alcohol or drug abuse within 12 months prior to screening
* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(s)
* History or evidence of any other clinically significant disorder, condition or disease that in the opinion of the Investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2012-11-07 (Actual); Primary Completion 2015-01-07 (Actual); Study Completion 2015-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (38):
- United States (9):
  - Research Site, Santa Monica, California
  - Research Site, Lakewood, Colorado
  - Research Site, Longmont, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Bethesda, Maryland
  - Research Site, Hagerstown, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, West Haverstraw, New York
  - Research Site, Houston, Texas
- Australia (6):
  - Research Site, Maroubra, New South Wales
  - Research Site, Penrith, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Box Hill, Victoria
  - Research Site, Geelong, Victoria
  - Research Site, Parkville, Victoria
- Belgium (8):
  - Research Site, Brussels
  - Research Site, Genk
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Merksem
  - Research Site, Tessenderlo
  - Research Site, Wilrijk
  - Research Site, Yvoir
- Canada (5):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Ballerup Municipality
  - Research Site, Vejle
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Torun
  - Research Site, Warsaw
- Spain (3):
  - Research Site, Granada, Andalusia
  - Research Site, Barcelona, Catalonia
  - Research Site, Madrid

REFERENCES:
- [Background] Miller PD, Pannacciulli N, Brown JP, Czerwinski E, Nedergaard BS, Bolognese MA, Malouf J, Bone HG, Reginster JY, Singer A, Wang C, Wagman RB, Cummings SR. Denosumab or Zoledronic Acid in Postmenopausal Women With Osteoporosis Previously Treated With Oral Bisphosphonates. J Clin Endocrinol Metab. 2016 Aug;101(8):3163-70. doi: 10.1210/jc.2016-1801. Epub 2016 Jun 6. PMID 27270237
- [Background] Miller PD, Pannacciulli N, Malouf-Sierra J, Singer A, Czerwinski E, Bone HG, Wang C, Huang S, Chines A, Lems W, Brown JP. Efficacy and safety of denosumab vs. bisphosphonates in postmenopausal women previously treated with oral bisphosphonates. Osteoporos Int. 2020 Jan;31(1):181-191. doi: 10.1007/s00198-019-05233-x. Epub 2019 Nov 28. PMID 31776637
- [Background] Chotiyarnwong P, McCloskey E, Eastell R, McClung MR, Gielen E, Gostage J, McDermott M, Chines A, Huang S, Cummings SR. A Pooled Analysis of Fall Incidence From Placebo-Controlled Trials of Denosumab. J Bone Miner Res. 2020 Jun;35(6):1014-1021. doi: 10.1002/jbmr.3972. Epub 2020 Apr 2. PMID 31999376
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 37 centers in Belgium, Denmark, Poland, Spain, Canada, United States of America, and Australia. The first participant enrolled on 07 November 2012 and the last participant enrolled on 15 January 2014.
Pre-assignment Details: Participants were randomized in a 1:1 allocation ratio to receive either denosumab or zoledronic acid. Randomization was stratified by screening serum type I collagen C-telopeptide (sCTX) values (< 0.3 ng/mL, 0.3 to 0.5 ng/mL).
Groups:
- Zoledronic Acid 5 mg Q12M: Participants received zoledronic acid 5 mg by intravenous infusion once every 12 months (Q12M) on Day 1 and placebo to denosumab by subcutaneous injection on Day 1 and at Month 6.
- Denosumab 60 mg Q6M: Participants received denosumab 60 mg subcutaneous injection once every 6 months (Q6M) for 12 months and placebo to zoledronic acid by intravenous infusion on Day 1.
Period: Overall Study
Arm/Group | Zoledronic Acid 5 mg Q12M | Denosumab 60 mg Q6M
Started | 322 | 321
Received Study Treatment | 320 | 320
Completed | 312 | 313
Not Completed | 10 | 8
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Decision by Sponsor | 2 | 2
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid 5 mg Q12M | Denosumab 60 mg Q6M | Total
Number analyzed (Participants) | 322 | 321 | 643
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (7.7) | 68.5 (7.1) | 69.0 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 322 | 321 | 643
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 314 | 309 | 623
  Asian | 4 | 5 | 9
  Other | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 0 | 1 | 1
  Multiple | 1 | 0 | 1
Screening serum CTX [Number; unit: participants]
  < 0.3 ng/mL | 242 | 239 | 481
  ≥ 0.3 ng/mL | 78 | 82 | 160
  Missing | 2 | 0 | 2
Lumbar Spine Bone Mineral Density (BMD) T-score [Mean (Standard Deviation); unit: T-score] — BMD was measured using dual-energy x-ray absorptiometry (DXA) of the lumbar spine. The T-score is a comparison of a person's bone density with that of a healthy 30-year-old of the same sex. Lower scores (more negative) mean lower bone density: A T-score of -2.5 or lower qualifies as osteoporosis and a T-score of -1.0 to -2.5 signifies osteopenia, meaning below-normal bone density without full osteoporosis.
  T-score | -2.64 (0.86) | -2.74 (0.83) | -2.69 (0.84)
Total Hip BMD T-score [Mean (Standard Deviation); unit: T-score] | -1.93 (0.80) | -1.93 (0.74) | -1.93 (0.77)
Femoral Neck BMD T-score [Mean (Standard Deviation); unit: T-score] | -2.17 (0.68) | -2.17 (0.66) | -2.17 (0.67)
Prior Oral Bisphosphonate Duration [Mean (Standard Deviation); unit: years] | 6.35 (3.68) | 6.21 (3.84) | 6.28 (3.76)
Historical Fractures [Number; unit: participants] — An osteoporotic fracture is defined as a reported fracture excluding skull fracture, facial bones fracture, fingers fracture and toes fracture, fractures with high trauma severity, and pathological fractures.
  participants
    Any prior fracture | 159 | 169 | 328
    Prior osteoporotic fracture | 121 | 120 | 241
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 24.31 (4.18) | 24.27 (3.99) | 24.29 (4.08)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density at Month 12 - Non-inferiority Analysis
Description: Bone mineral density (BMD) of the lumbar spine was measured by dual-energy x-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging facility.
Time Frame: Baseline and Month 12
Population: The primary efficacy analysis set includes all randomized participants who have a baseline BMD measurement and at least one postbaseline BMD measurement. Any postbaseline BMD value obtained at the early termination visit was carried forward as the month 12 value (ie, last observation carried forward [LOCF]).
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Zoledronic Acid 5 mg Q12M | Denosumab 60 mg Q6M
Number analyzed (Participants) | 312 | 314
percent change | 1.1 [0.7 to 1.5] | 3.2 [2.8 to 3.6]
Statistical Analysis 1: Comparison: Zoledronic Acid 5 mg Q12M vs Denosumab 60 mg Q6M; A step-down sequential testing procedure was used in order to maintain the overall type I error rate at 5% for the tests of primary and secondary BMD endpoints. For the non-inferiority analysis the 1-sided significance level was 2.5%; Test type: Non-Inferiority or Equivalence — The lower bound of the 2-sided 95% confidence interval (CI) of (denosumab - zoledronic acid) was compared with the non-inferiority margin of -0.46% for assessing non-inferiority; p < 0.0001, ANCOVA; The model included treatment, screening sCTX, baseline BMD, DXA machine type (Hologic or Lunar), and baseline BMD-by-machine type interaction; Treatment Difference = 2.1, 95% CI 2-sided [1.6 to 2.6] — Treatment difference = denosumab - zoledronic acid

2. Secondary Outcome: Percent Change From Baseline in Total Hip BMD at Month 12 - Non-inferiority Analysis
Description: BMD of the hip was measured by DXA. DXA scans were analyzed by a central imaging facility.
Time Frame: Baseline and Month 12
Population: The primary efficacy analysis set; any postbaseline BMD value obtained at the early termination visit was carried forward as the month 12 value (ie, LOCF).
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Zoledronic Acid 5 mg Q12M | Denosumab 60 mg Q6M
Number analyzed (Participants) | 309 | 311
percent change | 0.6 [0.3 to 0.8] | 1.9 [1.7 to 2.2]
Statistical Analysis 1: Comparison: Zoledronic Acid 5 mg Q12M vs Denosumab 60 mg Q6M; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The lower bound of the 2-sided 95% CI) of (denosumab - zoledronic acid) was compared with the non-inferiority margin of -0.51% for assessing non-inferiority; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 1.4, 95% CI 2-sided [1.0 to 1.7] — Treatment difference = denosumab - zoledronic acid

3. Secondary Outcome: Percent Change From Baseline in Lumbar Spine BMD at Month 12 - Superiority Analysis
Time Frame: Baseline and Month 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Zoledronic Acid 5 mg Q12M | Denosumab 60 mg Q6M
Number analyzed (Participants) | 312 | 314
percent change | 1.1 [0.7 to 1.5] | 3.2 [2.8 to 3.6]
Statistical Analysis 1: Comparison: Zoledronic Acid 5 mg Q12M vs Denosumab 60 mg Q6M; A step-down sequential testing procedure was used in order to maintain the overall type I error rate at 5% for the tests of primary and secondary BMD endpoints. For the superiority analysis the 2-sided significance level was 5%; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 2.1, 95% CI 2-sided [1.6 to 2.6] — Treatment difference = denosumab - zoledronic acid

4. Secondary Outcome: Percent Change From Baseline in Total Hip BMD at Month 12 - Superiority Analysis
Time Frame: Baseline and Month 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Zoledronic Acid 5 mg Q12M | Denosumab 60 mg Q6M
Number analyzed (Participants) | 309 | 311
percent change | 0.6 [0.3 to 0.8] | 1.9 [1.7 to 2.2]
Statistical Analysis 1: Comparison: Zoledronic Acid 5 mg Q12M vs Denosumab 60 mg Q6M; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 1.4, 95% CI 2-sided [1.0 to 1.7] — Treatment difference = denosumab - zoledronic acid

ADVERSE EVENTS:
Time Frame: 12 months
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Zoledronic Acid 5 mg Q12M | Denosumab 60 mg Q6M
Serious Adverse Events (participants affected / at risk) | 29/320 | 25/320
Other Adverse Events (participants affected / at risk) | 22/320 | 15/320
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 5 mg Q12M (N=320) | Denosumab 60 mg Q6M (N=320)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Drug interaction (General disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Vulval abscess (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 2
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral thrombosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Ischaemic stroke (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Knee operation (Surgical and medical procedures) | 1 | 0
Tendon operation (Surgical and medical procedures) | 0 | 1
Varicose vein operation (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 5 mg Q12M (N=320) | Denosumab 60 mg Q6M (N=320)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.